CLINICAL TRIAL: NCT02152059
Title: A Phase II Study of BIBF1120 in Recurrent and Platinum-Sensitive Small Cell Lung Cancer (SCLC)
Brief Title: A Study to Evaluate the Good and Bad Effects of BIBF1120 in Small Cell Lung Cancer Patients Who Have Previously Benefited From First-line Platinum-based Chemotherapy
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: contract issues
Sponsor: AHS Cancer Control Alberta (Other)
Collaborators: Cross Cancer Institute (Other); Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BIBF-SCLC-001
Record Dates: First submitted 2014-05-29; First posted 2014-06-02 (Estimated); Last update posted 2016-07-06 (Estimated); Status verified 2016-07

CONDITIONS: Small Cell Lung Cancer; Platinum-sensitive
Keywords: Small cell lung cancer; BIBF1120; nintedanib; platinum-sensitive
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — nintedanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BIBF1120 (Experimental): BIBF1120 200 mg twice daily continuously
  Interventions: Drug: BIBF1120

INTERVENTIONS:
Drug: BIBF1120 — BIBF1120 is a VEGFR, FGFR and PDGFR inhibitor
  Other Names: Nintedanib

SUMMARY:
This study is being done to evaluate the good and bad effects of BIBF1120 in recurrent, platinum-sensitive small cell lung cancer patients and to see if BIBF1120 may or may not be more effective and better tolerated than standard therapy.

The purpose of this study is to:

* Find out the proportion of patients with their small small cell lung cancer controlled for at least 90 days after treatment with BIBF1120
* Compare the response rate, survival and side effects of BIBF1120 in recurrent, platinum-sensitive small cell lung cancer patients
* Identify a group of patients who will benefit the most from BIBF1120 In this study, patients will receive BIBF1120 at 200 mg twice daily continuously. A cycle will be 21 days. During treatment, the dose of BIBF1120 will be held or reduced to lower doses if patients do not tolerate it well or if the doctors are concerned about the side effects of BIBF1120 on individual patients.

DETAILED DESCRIPTION:
This study is being done to evaluate the effects of BIBF1120 in recurrent, platinum-sensitive small cell lung cancer patients.

Primary Objectives:

* To investigate the efficacy and safety of a novel VEGFR-2 and FGFR-1 targeting agent, BIBF1120, in previously treated, platinum-sensitive small cell lung cancer patients.

Secondary Objectives:

* To correlate response to the apoptotic biomarkers, Bcl-XL/Bcl-2 and FDGR-1 amplification.
* To correlate response with baseline FLT-PET SUV uptake and change in FLT-PET SUV uptake.

All eligible patients will be treated with 200 mg bid of BIBF1120 daily and 21 days will be considered as one cycle

ELIGIBILITY:
Inclusion Criteria:

* Age > 18
* Recurrent and platinum-sensitive small cell lung cancer (SCLC): defined as those patients with SCLC recurrence at least 3 months from the last dose of platinum-based chemotherapy. Definition of platinum-sensitive disease is patient with at least 3 months of progression-free duration after finishing first-line platinum-based chemotherapy.
* Histological diagnosis of small cell lung cancer (including Oat cell carcinoma, small cell neuroendocrine tumor). Patients with archival tumor samples will be collected for further translational studies. For those who have no archival tumor samples, without due harm, a fresh biopsy can be obtained.
* As progression-free survival (PFS) or PFS rate is the endpoint, all patients enrolled must have measurable (per RECIST 1.1 Criteria) radiological progression of disease on radiological investigations.
* ECOG performance status of 0-2
* Adequate hematological function defined as hemoglobin > 90 g/L, ANC > 1500/uL and platelets > 100, 000/uL.
* Adequate renal function defined as creatinine < 1.5 x ULN or creatinine clearance > 45 mL/min (Cockcroft-Gault).
* Adequate liver function defined as AST/ALT < 1.5 x ULN or < 2.5 x ULN in the presence of liver metastases and total bilirubin < 1.5 x ULN.
* INR/PTT < 1.5 x ULN
* Left ventricular function by echocardiogram > institutional lower limit of normal.
* Women of childbearing potential and all must use adequate birth control. A serum pregnancy test must be performed within 72 hours from enrollment for all eligible women of childbearing potential.
* The absence of any significant psychiatric and medical condition that will potentially affect compliance to therapy or will be adversely affected by the experimental therapy.
* Able to swallow oral medication.
* Life expectancy of at least 12 weeks.
* All patients enrolled must have at least one prior platinum-based chemotherapy regimen in either the limited staged or extensive staged setting.
* All patients must have a blood pressure of 150/90 mm Hg or less at the time of enrollment. Patients who have been on anti-hypertensives will be eligible if their blood pressure is less than 150/90 mm Hg on enrollment with no increase of their anti-hypertensive medications for the 2 weeks prior to enrollment.
* Signed and dated written informed consent prior to enrollment in the study in accordance with ICH-GCP guidelines and to the local legislation.

Exclusion Criteria:

* Symptomatic, untreated brain metastasis. Patients with asymptomatic brain metastasis defined as those with no CNS symptoms, no concurrent significant edema on CT or MRI of the brain and no concurrent corticosteroid therapy will be eligible. Those with leptomeningeal disease will NEVER be eligible due to overall poor prognosis. Patients who have treated brain metastasis without concurrent corticosteroid and anti-convulsant therapy and without progression on CT or MRI scan of the brain for at least 60 days will be eligible
* Symptoms of congestive heart failure, myocardial infarction or angina within 6 months.
* Previous allergy to VEGR or FGF tyrosine kinase inhibitor.
* Current therapeutic coumadin treatment.
* History of pulmonary embolism, deep vein thrombosis within the past 1 year. Patients with any prior history of peripheral arterial thrombosis are not eligible.
* History of hemoptysis of more than 5 mL per episode or more than 10 mL/week in total within the past 3 months.
* History of bleeding disorder.
* Surgery, hormonal therapy, chemotherapy, radiation therapy or other investigational agents within 28 days of enrollment, with the exception of low dose palliative RT (20 Gy or less involving < 10% bone marrow).
* History of recent gastrointestinal bleeding, obstruction or perforation of malabsorption syndrome.
* History of QT c > 480 ms on ECG or hsitory of cardiac arrhythmia or treatment with anti-arrhythmic except for atrial fibrillation or any history of second- or third-degree heart block.
* Diagnosis of HIV infection or AIDS.
* Diagnosis of interstitial lung disease.
* Radiotherapy (except extremities) within the past 2 months prior to baseline imaging.
* Persistence of clinically relevant therapy-related toxicity from previous chemotherapy and/or radiotherapy.
* Leptomeningeal disease.
* Radiographic evidence of cavitary or necrotic tumors.
* Centrally located tumors with radiographic evidence (CT or MRI) of local invasion of major blood vessels. As small cell lung cancer is often presented as a mediastinal mass, compression of mediastinal blood vessels will be allowed.
* Therapeutic anticoagulation (except low-dose heparin and/or heparin flush as needed for maintenance of an in-dwelling intravenous device) or anti-platelet therapy (except for low-dose therapy with acetylsalicylic acid < 325 mg per day).
* Major injuries within the past 10 days prior to start of study treatment with incomplete wound healing and/or planned surgery during the on-treatment study period.
* History of clinically significant haemorrhagic or thromboembolic event in the past 6 months.
* Proteinuria CTCAE grade 2 or greater.
* Other malignancies within the past 5 years other than basal cell skin cancer or carcinoma in situ of the cervix.
* Active serious infections, in particular if requiring systemic antibiotic or antimicrobial therapy.
* Active or chronic hepatitis C and/or B infection.
* Patients who are sexually active and unwilling to use a medically acceptable method of contraception (e.g. such as implants, injectables, combined oral contraceptives, some intrauterine devices or vasectomised partner for participating females, condoms for participating males) during the trial and for at least 3 months after end of active therapy. Patients who are pregnant and/or lactating are not eligible.
* Active alcohol or drug abuse.
* Significant weight loss (> 10% of body weight) within past 6 months prior to inclusion into the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-07; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Disease control rate | 90 days

SECONDARY OUTCOMES:
Disease response rate | every 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Quincy Chu, MD, Principal Investigator — Alberta Health services
Locations (1):
- Cross Cancer Institute, Edmonton, Alberta, Canada